CLINICAL TRIAL: NCT00777192
Title: Prospective Study of Symptoms Related to Oxaliplatin-based Regimens in the Treatment of Colorectal Cancer
Brief Title: Longitudinal Study of Symptoms in Colorectal Cancer
Status: Terminated | Type: Observational
Why Stopped: Terminated at continuing review
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007-0637
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; Cancers of the colon and rectum; Oxaliplatin; oxaliplatin chemotherapy; inflammatory cytokines; neurocognitive symptoms; neuropsychiatric symptoms
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and cell samples will also be collected during chemotherapy for analysis of cytokines and their relationship to symptom production.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptoms in Colorectal Cancer: Colorectal Cancer Patients Receiving Oxaliplatin Chemotherapy
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — 20 Minute Questionnaires beginning Visit 1, to measure pain/other symptoms, mood, and quality of life

SUMMARY:
The goal of this research study is to learn more about the pain and/or other symptoms that patients may experience within five years from CRC diagnosis. Researchers also want to learn how genetic differences may affect the symptoms patients experience from cancer and cancer therapy.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete 5 questionnaires during a regularly scheduled visit. The questionnaires are designed to measure pain and other symptoms, your mood, and your quality of life.

You will also give a tissue sample by inserting a cotton tipped swab into your mouth and rubbing firmly against the inside of your cheek or underneath your lower or upper lip for about 1 minute at the most.

Completing the 5 questionnaires and the swab sample should take about 30 minutes.

Length of Study:

After you complete the questionnaires and the swab sample collection, your active participation in this study will be over.

This is an investigational study.

Up to 500 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with colorectal cancer meeting one of the following criteria: 1. naive to oxaliplatin or to any microtubule stabilizing agents (e.g. Taxol, Abraxane, Ixabepilone) but scheduled for combined oxaliplatine chemotherapy (longitudinal study cohort 1); or 2. during first 5 years from colorectal cancer diagnosis (cross-sectional study cohort). This second cohort may include patients with colorectal cancer from the original 12-month study (the longitudinal cohort), both those who completed the study and those who dropped out. It may also include new patients who did not participate in the longitudinal phase of the study.
2. Patients >= 18 years old.
3. Patients who speak English or Spanish.

Exclusion Criteria:

1. Cohort 1 patients with a neuropathy score of 1 or greater on the NCI's Common Terminology Criteria (CTCv3.0).
2. Patients who do not understand the intent of the study.
3. Cohort 1 patients unable to use the interactive voice response (IVR) system due to physical limitations (e.g., hearing impairment).
4. Cohort 1 patients with a history of inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having oxaliplatin chemotherapy as a treatment for colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Association between inflammatory cytokines and development of treatment-related symptom burden in colorectal cancer patients | 5 Years

SECONDARY OUTCOMES:
Primary afferent function in colorectal cancer patients receiving chemotherapy by quantitative sensory testing over time | 5 Years
Neurocognitive and neuropsychiatric symptoms in colorectal cancer patients | Neuropsychological test battery at baseline and 3 + 6 month follow ups

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD. MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wang XS, Shi Q, Dougherty PM, Eng C, Mendoza TR, Williams LA, Fogelman DR, Cleeland CS. Prechemotherapy Touch Sensation Deficits Predict Oxaliplatin-Induced Neuropathy in Patients with Colorectal Cancer. Oncology. 2016;90(3):127-35. doi: 10.1159/000443377. Epub 2016 Feb 17. PMID 26882477
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org